CLINICAL TRIAL: NCT05662449
Title: A Cohort Study of Bioabsorbable Screws for Syndesmosis Fixation in Ankle Fracture
Brief Title: A Cohort Study of Bioabsorbable Screws for Syndesmosis Fixation Fixation in Ankle Fracture
Acronym: Synfix
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NHS Grampian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 209339
Record Dates: First submitted 2021-03-08; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Syndesmotic Injuries; Ankle Fractures; Ankle Injuries and Disorders
MeSH Terms: conditions — Ankle Injuries; Ankle Fractures; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ankle fracture with syndesmosis injury: Syndesmosis fixation using bioabsorbable screw
  Interventions: Device: Syndesmosis fixation using Activascrew

INTERVENTIONS:
Device: Syndesmosis fixation using Activascrew — as described prior

SUMMARY:
The investigators aim to evaluate the fixation of the ankle syndesmosis in appropriate ankle fractures with bioabsorbable screws.

Ankle fractures are common, and a proportion of them involve both fracture of the bone and also disruption of the syndesmosis, a strong ligamentous complex connecting the distal fibula and tibia. If left without fixation this causes a high incidence of pain and early arthritis. The most common technique for fixation of this syndesmosis involves the use of the same type of metal screws used to fix the fractured bones. As the syndesmosis permits small degrees of movement in normal subjects, fixation of this with metal usually leads to screw breakage and, or pain. It is common practice to remove these screws after a period of time once the syndesmosis has healed in the correct position.

Bioabsorbable screws have the advantage of allowing small increments of movement, and also resorb naturally therefore do not have to be removed with a second surgical procedure. They are used in other centres worldwide, and the investigators therefore seek to evaluate syndesmosis fixation with them in their unit. The investigators would aim to recruit patients who have a syndesmotic injury requiring fixation, and who can consent to participating. They would undergo an identical surgical procedure to the standard current practice, apart from using a bioabsorbable screw in exchange for the metallic screw for syndesmosis fixation. All other components would remain unchanged, as would post operative protocol and management. To evaluate the fixation the investigators would use a limited CT scan (equivalent of about 3 months background radiation) after the time of fixation and at one year. This will help to assess the maintenance of reduction of the syndesmosis with time. The investigators would also assess patient reported outcome measures and pain scores, length of procedure and intraoperative radiation levels, weight bearing distribution tests, as well as any complication that may arise.

DETAILED DESCRIPTION:
Surgical Technique The operation requires the patient positioned supine with a sandbag beneath the ipsilateral buttock to internally rotate the leg to permit the ankle and foot to sit in neutral. Appropriate antibiotics as per local guidelines should be administered prior to insufflation of a tourniquet. Fluoroscopy is required throughout the procedure and should be positioned on the contralateral side to the injured limb to improve the access for the surgical team.

Depending on the injury type the fibula may or may not require fixation (maissoneuve or weber B/C type injury). This will be performed if necessary via a direct lateral approach to the fibula, and fixation as per surgeon preference appropriate for the fracture configuration. Typically a lag screw and one-third tubular neutralisation plate is used. Plates should be applied to the posterolateral surface of the fibula to permit passage of the syndesmosis screw through the plate and for increased mechanical stability. Following this the syndesmosis will be reduced with the foot plantigrade using large pointed reduction forceps with or without a K-wire. Medial malleolar fixation, if required, is performed after fibula fixation.

Bio-absorbable screw fixation A single 4.5 mm fully threaded ActivascrewTM (2094913CE01) is placed through four cortices if the fibula fracture is being fixed, through the plate if feasible. Two are used in the case of high fibula or maissoneuve injuries. These will all be through four cortices. A countersink may be used. The screws should be placed parallel to the tibial plafond, 2-4cm proximal to the tibio-talar joint and 30° from posterior to anterior. In the case of fibula fixation this should be though the plate if feasible. The reduction of the syndesmosis and appropriate placement of the positioning screw(s) should be checked intra-operatively with fluoroscopy. The syndesmosis is reduced, using reduction forceps. A hole is drilled with the 3.5mm drill, then tapped with the 4.5mm tap and measured. The ActivascrewTM holder and screwdriver are used to pick up and insert the desired screw. Once the screw is in position the insertion adapter is removed and discarded.

Standardised rehabilitation protocol Post operatively the patient remains non weight-bearing in a Plaster for a total of 6 weeks with a cast change, wound check and removal of sutures at 2 weeks. Following this the patient would then remain partial weight bearing in a protective boot for a further 6 weeks. The patients should be prescribed 6 weeks of Low Molecular Weight Heparin for venous thromboembolic prophylaxis as per local protocol.

Sample size considerations A total number of 40 patients should be sufficient to assess the outcome of fixation using this device.

Patients selection and enrolment Patients will be thoroughly screened to assess their suitability for the study and must fit the inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* • Patient has a Weber C fibula fracture with or without a medial malleolus fracture and evidence of radiological syndesmotic widening on intra-operative stressing

  * Patient has a Weber B fracture with evidence of syndesmosis widening radiologically on stressing intra-operatively
  * Patient has a maissoneuve type injury with evidence of syndesmotic diastasis
  * Patient mobilises independently, with or without aids.
  * Patient has given formal consent to be involved in the trial and has completed the study consent form
  * Patient is likely to comply with study requirements
  * Patient is over the age of 18 years and under 65 years

Exclusion Criteria:

* • Immobility

  * Presence of a posterior malleolus fracture involving >25% of articular surface
  * Open fractures
  * Pathological fractures
  * Other fractures involving the same lower extremity
  * Patient unwilling to give informed consent to be included in the trial
  * Patient has other injuries that would influence the study
  * Any ankle fracture that the treating surgeon feels inappropriate to be included in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Meets above criteria with appropriate ankle fracture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Computerised Tomography (CT) scan syndesmosis | Change in reduction between 2 weeks and 1 year post operatively
  All patients will undergo focused CT scanning two weeks post operatively and at one year. A customised foot holding device will enable to scan to be taken with both feet in neutral alignment (Evolution supine foot positioner, Vasocare Ltd). Assessment will be made in comparison with the contralateral side to assess reduction of the syndesmosis. Quantitive measurement of reduction will be measured using an established technique from the paper cited below in references.

SECONDARY OUTCOMES:
Surgical Duration | Intraoperative
  Tourniquet time (minutes) to represent this
X- Ray (XR) Radiation exposure time and total dose | Intraoperative
  Image intensifier screening total time(seconds) and dose(cGycm2)
Olerud-Molander Ankle Score (OMAS) | Pre-operative (baseline), 3 months, 6 months and 1 year post operatively. Absolute values measured as well as change in score over time intervals noted.
  (Olerud-Molander Ankle Scores). Verified and reproducible patient reported scale for ankle function and symptoms. Range 0-100. High score is better.
EQ5D3L (European Quality of Life 5 Dimensions 3 Level Version) | Pre-operative (baseline), 3 months, 6 months and 1 year post operatively.Absolute values measured as well as change in score over time intervals noted.
  EQ-5D-3L (European Quality of Life 5 Dimensions 3 Level Version). Validated patient health questionnaire. Score range 5-15. Lower score is better.
EQ-5D-3L VAS (European Quality of Life 5 Dimensions 3 Level Version) Health state | Pre-operative (baseline), 3 months, 6 months and 1 year post operatively.Absolute values measured as well as change in score over time intervals noted.
  Validated patient health questionnaire. Score range 0-100. High score is better.
American Academy Orthopaedic Surgeons Foot and Ankle Outcomes (AAOSFA) | Pre-operative (baseline), 3 months, 6 months and 1 year post operatively.Absolute values measured as well as change in score over time intervals noted.
  Verified and reproducible patient reported scale for Pain, Function, Shoe wear and Alignment (numerical scoring system). Range 0-100. High score is better.
Complications | Up to 12 months
  Details of any recorded minor and major complications
X-Rays (XR) | 2 weeks, 6 weeks, 3 months, 6 months and 1 year post operatively.
  Mortise and lateral XR to assess alignment if satisfactory
Weight bearing tests | 3 months, 6 months and 1 year post operatively
  Assessment if can weight bearing. Stand on two sets of scales, one foot on each scale. Timed over 1 minute and assess how much weight (kg) is on each scale at 15 second intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Johnstone, MBChB FRCS, Principal Investigator — NHS Grampian
Locations (1):
- Aberdeen Royal Infirmary, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Phisitkul P, Ebinger T, Goetz J, Vaseenon T, Marsh JL. Forceps reduction of the syndesmosis in rotational ankle fractures: a cadaveric study. J Bone Joint Surg Am. 2012 Dec 19;94(24):2256-61. doi: 10.2106/JBJS.K.01726. PMID 23318616

DOCUMENTS (2):
  • Study Protocol (2022-07-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT05662449/Prot_000.pdf
  • Informed Consent Form (2020-10-25): https://cdn.clinicaltrials.gov/large-docs/49/NCT05662449/ICF_001.pdf